CLINICAL TRIAL: NCT02643992
Title: Per-procedural Concentration of Direct Oral Anticoagulants
Acronym: CORIDA
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGR_2014-13
Record Dates: First submitted 2015-12-30; First posted 2015-12-31 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Per-procedural Concentrations of Oral Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: DOAC concentration measurement

SUMMARY:
Background: Peri-procedural management of direct oral anticoagulants (DOAC) is challenging. The optimal duration of pre-procedural discontinuation that guarantees a minimal DOAC concentration ([DOAC]) at surgery is unknown. The usual 48-hour discontinuation might not be sufficient for all patients.

Objectives: To investigate the factors associated with per-procedural [DOAC]. To test the hypothesis that a 48-hour DOAC discontinuation is not sufficient to ensure a minimal perprocedural [DOAC], defined as [DOAC] < 30 ng/mL.

Methods: Patients treated with DOAC, and requiring any invasive procedure will be included in this multicentre, prospective, observational study. [DOAC], will be measured during invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years-old
* undergoing invasive procedure
* treated with DOAC

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing invasive procedure and treated with DOAC
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
DOAC concentration | beginning of invasive procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris, France

REFERENCES:
- [Derived] Godier A, Martin AC, Lessire S, Mullier F, Leblanc I, Gouin-Thibault I. Concentrations of direct oral anticoagulants according to guidelines for the periprocedural management of low bleeding risk procedures. Anaesth Crit Care Pain Med. 2020 Feb;39(1):121-122. doi: 10.1016/j.accpm.2019.04.004. Epub 2019 Apr 13. No abstract available. PMID 30991108